CLINICAL TRIAL: NCT03009123
Title: Erectile Dysfunction and the Future Risk of Prostate Cancer: a Population-based Longitudinal Follow-up Study With Concurrent Double Comparison Cohorts
Brief Title: Will Erectile Dysfunction Increase the Risk of Prostate Cancer
Acronym: EDtoPC
Status: Completed | Type: Observational
Sponsor: Kuang Tien General Hospital (Other)
Collaborators: Asia University (Other); National Central University, Taiwan (Other)
Responsible Party: Principal Investigator, Victor C. Kok, MMedSc, MD, PhD, FACP, Ass. Professor, Kuang Tien General Hospital
Other Study IDs: KTGH-ASIAU-obs-erectile
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Erectile Dysfunction
Keywords: cohort study; prostate cancer; population-based study; benign prostatic hypertrophy
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Erectile dysfunction group: Group contains men with physician-diagnosed erectile dysfunction
  Interventions: Other: Erectile dysfunction
- General population men without ED: Men 50 years and older having no ED and pre-existing prostate cancer
- Symptomatic BPH group without ED: Men 50 years old older with symptomatic prostatic hypertrophy but with no ED nor pre-existing prostate cancer

INTERVENTIONS:
Other: Erectile dysfunction — Patients with ED are considered belonging to the exposure group.
  Groups: Erectile dysfunction group

SUMMARY:
The rationale for investigating the hypothesis that there is an association between erectile dysfunction (ED) and the subsequent development of prostate cancer is based on three assumptions: 1) baseline ED is common in most if not all of the cross-sectional studies in men with prostate cancer; 2) the development of ED and prostate cancer may have certain shared common risk factors; and 3) the use of testosterone for the treatment of ED has been suspected to be associated with prostate cancer development. Controversy exists over whether men with ED have an increased risk of subsequent prostate cancer. Few studies have evaluated the risk of developing prostate cancer for men with ED. The investigators, therefore, conducted a population-based longitudinal study with eight years' follow-up to examine this association and to evaluate the magnitude of the risk.

ELIGIBILITY:
Inclusion Criteria:

* men 50 years and older with no pre-existing prostate cancer

Exclusion Criteria:

* less than 50 years old
* pre-existing prostate cancer

Ages: 50 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort was constructed from the Taiwan National Health Insurance Research Dataset. From among men with no pre-existing prostate cancer, we formed an ED group of men ≥50 years of age and a non-ED general population comparison group of men matched 1:4 by age and index date of the ED group and a concurrent second comparison group of men older than 50 with benign prostatic hypertrophy.
Sampling Method: Non-Probability Sample
Enrollment: 21558 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-15 (Actual); Study Completion 2017-05-06 (Actual)

PRIMARY OUTCOMES:
Incident prostate cancer | through study completion, up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Victor C Kok, MD, PhD, Study Director — Disease Informatics Research Unit, Asia University Taiwan
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sairam K, Kulinskaya E, Boustead GB, Hanbury DC, McNicholas TA. Prevalence of undiagnosed prostate cancer in men with erectile dysfunction. BJU Int. 2002 Feb;89(3):261-3. doi: 10.1046/j.1464-4096.2001.01271.x. PMID 11856107
- [Background] Saitz TR, Serefoglu EC, Trost LW, Thomas R, Hellstrom WJ. The pre-treatment prevalence and types of sexual dysfunction among patients diagnosed with prostate cancer. Andrology. 2013 Nov;1(6):859-63. doi: 10.1111/j.2047-2927.2013.00137.x. Epub 2013 Oct 11. PMID 24127273
- [Background] Resnick MJ, Barocas DA, Morgans AK, Phillips SE, Chen VW, Cooperberg MR, Goodman M, Greenfield S, Hamilton AS, Hoffman KE, Kaplan SH, Paddock LE, Stroup AM, Wu XC, Koyama T, Penson DF. Contemporary prevalence of pretreatment urinary, sexual, hormonal, and bowel dysfunction: Defining the population at risk for harms of prostate cancer treatment. Cancer. 2014 Apr 15;120(8):1263-71. doi: 10.1002/cncr.28563. Epub 2014 Feb 7. PMID 24510400
- [Background] Chou PS, Chou WP, Chen MC, Lai CL, Wen YC, Yeh KC, Chang WP, Chou YH. Newly diagnosed erectile dysfunction and risk of depression: a population-based 5-year follow-up study in Taiwan. J Sex Med. 2015 Mar;12(3):804-12. doi: 10.1111/jsm.12792. Epub 2014 Dec 5. PMID 25475605
- [Background] Lee PH, Kok VC, Chou PL, Ku MC, Chen YC, Horng JT. Risk and clinical predictors of osteoporotic fracture in East Asian patients with chronic obstructive pulmonary disease: a population-based cohort study. PeerJ. 2016 Oct 27;4:e2634. doi: 10.7717/peerj.2634. eCollection 2016. PMID 27812429
- [Background] Kok VC, Horng JT, Hung GD, Xu JL, Hung TW, Chen YC, Chen CL. Risk of Autoimmune Disease in Adults with Chronic Insomnia Requiring Sleep-Inducing Pills: A Population-Based Longitudinal Study. J Gen Intern Med. 2016 Sep;31(9):1019-26. doi: 10.1007/s11606-016-3717-z. Epub 2016 Apr 29. PMID 27130621
- [Background] Kok VC, Sung FC, Kao CH, Lin CC, Tseng CH. Cancer risk in East Asian patients associated with acquired haemolytic anaemia: a nationwide population-based cohort study. BMC Cancer. 2016 Feb 4;16:57. doi: 10.1186/s12885-016-2098-3. PMID 26846920
- [Background] Kok VC, Tsai HJ, Su CF, Lee CK. The Risks for Ovarian, Endometrial, Breast, Colorectal, and Other Cancers in Women With Newly Diagnosed Endometriosis or Adenomyosis: A Population-Based Study. Int J Gynecol Cancer. 2015 Jul;25(6):968-76. doi: 10.1097/IGC.0000000000000454. PMID 25893280
- [Background] Kok VC, Horng JT, Huang HK, Chao TM, Hong YF. Regular inhaled corticosteroids in adult-onset asthma and the risk for future cancer: a population-based cohort study with proper person-time analysis. Ther Clin Risk Manag. 2015 Mar 26;11:489-99. doi: 10.2147/TCRM.S80793. eCollection 2015. PMID 25848295
- [Background] Kok VC, Horng JT, Huang JL, Yeh KW, Gau JJ, Chang CW, Zhuang LZ. Population-based cohort study on the risk of malignancy in East Asian children with juvenile idiopathic arthritis. BMC Cancer. 2014 Aug 29;14:634. doi: 10.1186/1471-2407-14-634. PMID 25174953
- [Background] Kok VC, Horng JT, Chang WS, Hong YF, Chang TH. Allopurinol therapy in gout patients does not associate with beneficial cardiovascular outcomes: a population-based matched-cohort study. PLoS One. 2014 Jun 4;9(6):e99102. doi: 10.1371/journal.pone.0099102. eCollection 2014. PMID 24897240
- [Background] Kok VC, Horng JT, Lin HL, Chen YC, Chen YJ, Cheng KF. Gout and subsequent increased risk of cardiovascular mortality in non-diabetics aged 50 and above: a population-based cohort study in Taiwan. BMC Cardiovasc Disord. 2012 Nov 21;12:108. doi: 10.1186/1471-2261-12-108. PMID 23170782